CLINICAL TRIAL: NCT01438346
Title: A Pilot Study of Two Group-based Intervention Programs for Patients With Substance Abuse Problems
Brief Title: Behavioral Treatment for Substance Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Yoshio Nakamura, Research Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00027696
Record Dates: First submitted 2011-09-16; First posted 2011-09-22 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Substance-Related Disorders
Keywords: Substance Abuse; Substance Addiction; Substance Dependence; Treatment program
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Substance Abuse Education (SED) (Active Comparator): The Substance Abuse Education (SED) group will serve as the control intervention in which participants will receive instruction on a variety of topics included in the substance abuse treatment program curriculum. These will include, but are not limited to, information about anger management, smoking cessation, women's issues, and stress management, and approaches to help reduce cravings. Each week the TAU group will meet and a House of Hope (HOH) clinical staff member will discuss the above and related issues and how these may help individuals deal with their substance abuse and related psychological issues.
  Interventions: Behavioral: Substance Abuse Education
- Mind-body Bridging (MBB) (Experimental): Participants in the experimental Mind-Body Bridging (MBB) group, in addition to their usual treatment for substance abuse, will additionally receive instruction on the basics of MBB, and will learn MBB techniques to help deal with their cravings and comorbid psychological conditions. A workbook will be incorporated into the curriculum to provide MBB participants with daily exercises and activities to help facilitate adherence to the MBB program.
  Interventions: Behavioral: Mind-body Bridging

INTERVENTIONS:
Behavioral: Substance Abuse Education — 10 weeks of usual care for substance abuse.
  Other Names: Substance abuse usual care; Substance abuse treatment as usual
  Arms: Substance Abuse Education (SED)
Behavioral: Mind-body Bridging — Two sessions per week for 10 weeks, besides usual care treatment for substance abuse.
  Other Names: Mind and Body Bridging Program
  Arms: Mind-body Bridging (MBB)

SUMMARY:
This pilot project will evaluate a new mind-body intervention called Mind-Body Bridging (MBB) for reducing substance abuse problems in women who are undergoing a substance abuse treatment program. The main hypothesis is that MBB will be more effective than the control (standard) intervention program in helping people reduce their craving for illicit substances and/or alcohol.

DETAILED DESCRIPTION:
This is a randomized clinical pilot study in which MBB will be compared with a standard treatment program for substance abuse. Both groups will run concurrently over the course of a 10-week period, twice per week.

ELIGIBILITY:
Inclusion Criteria:

* Substance abuse or dependence
* Resident/day client in the House of Hope substance abuse treatment program
* Minimum stay in treatment at House of Hope for 3.5 months
* Fluent in English

Exclusion Criteria:

* Psychosis
* Suicide risk
* Dementia
* Significant withdrawal risk
* Severe, unstable depression
* Requires intensive mental health treatment
* Cognitive impairment

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the measure of the Penn Alcohol and Craving Scale | Week 5 and Week 11
  Change from baseline in the extent of drug and alcohol craving at Week 5 and Week 11, as measured by a modified version of the Penn Alcohol and Craving Scale
Change from baseline in Alcohol and Drug Use Consequences Scale | Week 5 and Week 11
  Change from baseline in the measure of alcohol and drug consequences at Week 5 and Week 11, as measured by Alcohol and Drug Use Consequences Scale

SECONDARY OUTCOMES:
Subjective distress | Pre (Baseline) Mid (Week 5), Post (Week 11)
  Impact of Events Scale - Revised (IES-R) is a 22-item self-report measure that assesses subjective distress caused by traumatic events. The IES-R yields a total score (ranging from 0 to 88) and subscale scores can also be calculated for the Intrusion, Avoidance, and Hyperarousal subscales.
Depression | Pre (Baseline) Mid (Week 5), Post (Week 11)
  The Center for Epidemiologic Studies Depression Scale is one of the most common screening tests to determine an individual's depression quotient. The test measures depressive feelings and behaviors during the past week.
Sleep | Pre (Baseline) Mid (Week 5), Post (Week 11)
  The Medical Outcomes Study Sleep Scale (MOS-SS) provides an index of sleep problems and incorporates six sleep scale scores: 1) sleep disturbance, 2) sleep adequacy, 3) daytime somnolence, 4) snoring, 5) waking up short of breath with a headache, and 6) quantity of sleep. The MOS-SS is similar to the Pittsburgh Sleep Quality Index (PSQI) developed at the same time, which includes more questions about sleep disturbance with seven more items overall. The 1-week assessment is adapted from the normal 4-week retrospective assessment.
Mindfulness | Pre (Baseline) Mid (Week 5), Post (Week 11)
  The Five-facet Mindfulness Questionnaire (FFMQ) comprises five clear, interpretable facets of mindfulness: acting with awareness, observing, describing, non-judging, non-reacting.
Self-Compassion | Pre (Baseline) Mid (Week 5), Post (Week 11)
  Self compassion is measured by the Self-Compassion Scale that comprises 26 items. Self-compassion is an emotionally positive self-attitude that should protect against the negative consequences of self-judgment, isolation, and rumination (such as depression).
Well-being | Weekly for 11 weeks
  The Well-Being Index (WBI)is a 5-item scale developed and validated by the World Health Organization Collaborating Centre in Mental Health. The WBI will be used to assess whether participants show any changes in general well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshi Nakamura, Ph.D., Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - House of Hope, Salt Lake City, Utah
  - Pain Research Center, Anesthesiology, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No